CLINICAL TRIAL: NCT00840476
Title: A Two-way Crossover, Open-label, Single-dose, Fasting, Bioequivalence Study of Meloxicam 15 mg Tablets Versus Mobic® 15 mg Tablets in Normal Healthy Non-Smoking Male and Female Subjects
Brief Title: Meloxicam 15 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2824
Record Dates: First submitted 2009-02-06; First posted 2009-02-10 (Estimated); Results first posted 2009-08-04 (Estimated); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Meloxicam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Meloxicam (Experimental): Meloxicam 15 mg Tablet (test) dosed in first period followed by Mobic® 15 mg Tablet (reference) dosed in second period
  Interventions: Drug: Meloxicam 15 mg Tablets
- Mobic® (Active Comparator): Mobic® 15 mg Tablet (reference) dosed in first period followed by Meloxicam 15 mg Tablet (test) dosed in second period
  Interventions: Drug: Mobic® 15 mg Tablets

INTERVENTIONS:
Drug: Meloxicam 15 mg Tablets — 1 x 15 mg, single-dose fasting
  Arms: Meloxicam
Drug: Mobic® 15 mg Tablets — 1 x 15 mg, single-dose fasting
  Arms: Mobic®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of meloxicam from a test formulation Meloxicam 15 mg Tablets versus the reference Mobic® 15 mg Tablets under fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA bioequivalence statistical methods

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking male or female with a minimum age of 18 years (i.e. non-smoker or non tobacco user for at least 90 days prior to pre-study medical).
* Body mass Index (BMI = weight/height²) greater than or equal to 18.5 kg/m² and less than or equal to 29.9 kg/m².
* Availability of subject for the entire study period and willingness to adhere to protocol requirements, as evidenced by a signed Informed Consent Form.
* Normal findings in the physical examination, 12-lead ECG and vital signs (blood pressure between 100-140/60-90 mmHg, heart rate between 50-99 beats/min, temperature between 35.8ºC and 37.5ºC).
* Negative for drugs of abuse, nicotine, alcohol, hepatitis B-surface antigen, hepatitis C and HIV, and for female subjects, pregnancy (serum ß-CG).
* No clinical laboratory values outside of the acceptable range as defined by BCR, unless the Principal Investigator decides they are not clinically significant.
* Female subjects who are surgically sterile for at least six months or post-menopausal for at least one year, or who will avoid pregnancy prior to the study, during the study and up until one month after the end of the study.

Exclusion Criteria:

* Known history of hypersensitivity to meloxicam (for example Mobic®), or related drugs such as any other non-steroidal anti-inflammatory drugs (NSAID) such as acetylsalicyclic acid (e.g. Excedrin®, Aspirin®), ibuprofen (e.g. Motrin®), celecoxib (e.g. Celebrex®), Feldene®, Indocin®, Naprosyn®, Vioxx®, Toradol®, Clinoril®, Tolectin®, or Lodine®.
* Known history or presence of cardiac, pulmonary, gastrointestinal, endocrine, musculoskeletal, neurological, hematological, or liver disease, unless judged not clinically significant by the Principal Investigator, or medical designate.
* Any history or presence of peptic ulcer disease, gastrointestinal bleeding, or kidney disease.
* Known history or presence of food allergies, or any condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
* Any clinically significant illness during the last four weeks prior to entry into this study.
* Presence of any significant physical or organ abnormality.
* Any subject with history of drug abuse.
* Any psychiatric or psychological disease (including depression) unless deemed not clinically significant by the Principal Investigator, or medical designate.
* Use of any prescription medication within 14 days preceding entry into this study.
* Use of over-the-counter (OTC) medication within seven days preceding entry into this study (except for spermicidal/barrier contraceptive products).
* Female subjects: use of oral contraceptives or contraceptive implants (such as Norplant®) within 30 days prior to drug administration or a depot injection of progestogen drug (e.g. Depo-Provera®) within one year prior to drug administration.
* Female subjects: presence of pregnancy or lactation.
* Female subjects at risk of becoming pregnant must consent to using two medically acceptable methods of contraception throughout the entire study, including the washout period and for one month after the completion of the study. Medically acceptable barrier methods of contraception that may be used by the subject and/or partner include diaphragm with spermicide, IUD, condom with foam, and vaginal spermicidal suppository. Complete abstinence can be used alone as a method of contraception.
* Any subject who has had blood drawn within 56 days preceding this study, taken during the conduct of any clinical study at a facility other than BCR or within the lockout period specified by a previous study conducted at BCR.
* Participation in a clinical trial with an investigational drug within 30 days preceding this study.
* Any subject who has donated blood within 56 days preceding this study.
* Any subject who has participated as a plasma donor in a plasmapheresis program within seven days preceding this study.
* Any subject with a recent (less than one year) history of alcohol abuse.
* Significant or recent history of asthma (after 12 years of age), or familial history of asthma or aspirin-sensitive asthma, sever bronchospasm, nasal polyps or chronic sinusitis.
* Intolerance to venipuncture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2004-02; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Y. Tam, M.D., Principal Investigator — Biovail Contract Research
Locations (1):
- Biovail Contract Research, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Meloxicam (Test) First: Meloxicam 15 mg Tablet (test) dosed in first period followed by Mobic® 15 mg Tablet (reference) dosed in second period
- Mobic® (Reference) First: Mobic® 15 mg Tablet (reference) dosed in first period followed by Meloxicam 15 mg Tablet (test) dosed in second period
Period: First Intervention
Arm/Group | Meloxicam (Test) First | Mobic® (Reference) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Washout: 14 Days
Arm/Group | Meloxicam (Test) First | Mobic® (Reference) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Meloxicam (Test) First | Mobic® (Reference) First
Started | 14 | 14
Completed | 14 | 14
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Meloxicam (Test) First | Mobic® (Reference) First | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 14 | 27
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 4 | 12
  Male | 6 | 10 | 16
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 9 | 9 | 18
  Black | 3 | 4 | 7
  Asian | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Canada | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Cmax - Maximum Observed Concentration
Description: Bioequivalence based on Cmax
Time Frame: Blood samples collected over 96 hour period
Population: The data from two completed subjects was not included in the statistical analysis due to pre-dose concentrations greater than 5% of the individuals Cmax value.
Measure: Mean (Standard Deviation); unit: µg/mL
Groups:
- Meloxicam: Meloxicam 15 mg Tablet (test) dosed in either period
- Mobic®: Mobic® 15 mg Tablet (reference) dosed in either period
Arm/Group | Meloxicam | Mobic®
Number analyzed (Participants) | 26 | 26
µg/mL | 1.50 (0.41) | 1.51 (0.44)
Statistical Analysis 1: Comparison: Meloxicam vs Mobic®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 100.26, 90% CI [93.12 to 107.95] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

2. Primary Outcome: AUC0-inf - Area Under the Concentration-time Curve From Time Zero to Infinity (Extrapolated)
Description: Bioequivalence based on AUC0-inf
Time Frame: Blood samples collected over 96 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Meloxicam | Mobic®
Number analyzed (Participants) | 26 | 26
µg*h/mL | 46.89 (17.19) | 44.82 (16.83)
Statistical Analysis 1: Comparison: Meloxicam vs Mobic®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 105.14, 90% CI [100.27 to 110.25] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

3. Primary Outcome: AUC0-t - Area Under the Concentration-time Curve From Time Zero to Time of Last Non-zero Concentration (Per Participant)
Description: Bioequivalence based on AUC0-t
Time Frame: Blood samples collected over 96 hour period
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: µg*h/mL
Arm/Group | Meloxicam | Mobic®
Number analyzed (Participants) | 26 | 26
µg*h/mL | 43.25 (14.27) | 41.98 (15.42)
Statistical Analysis 1: Comparison: Meloxicam vs Mobic®; Test type: Non-Inferiority or Equivalence — Analysis of variance (ANOVA) was performed on pharmacokinetic parameters of AUC0-t, AUCinf and Cmax; Test/Ref Ratio of LS Means x 100 = 104.33, 90% CI [99.16 to 109.76] — Bioequivalence is established when 90% Confidence Interval falls within 80-125

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator is not permitted to discuss or publish trial results.